CLINICAL TRIAL: NCT00320567
Title: The Effect of Ortho Tri-Cyclen on Bone Mineral Density in Pediatric Subjects With Anorexia Nervosa: A Double-Blind, Placebo-Controlled Study
Brief Title: The Effect of Norgestimate/Ethinyl Estradiol on Bone Density in Pediatric Subjects With Anorexia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR008332
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Osteoporosis
Keywords: osteoporosis; anorexia nervosa; pediatric
MeSH Terms: conditions — Osteoporosis; Anorexia Nervosa | interventions — Moxifloxacin

ARMS (1):
- 001 (Experimental): norgestimate/ethinyl estradiol
  Interventions: Drug: norgestimate/ethinyl estradiol

INTERVENTIONS:
Drug: norgestimate/ethinyl estradiol

SUMMARY:
The purpose of this study is to evaluate the effect of norgestimate/ethinyl estradiol on lumbar spine (L1-L4) and total hip bone mineral density (BMD) in pediatric subjects with anorexia nervosa.

DETAILED DESCRIPTION:
Although oral contraceptives are prescribed in an effort to prevent bone loss in adolescents with anorexia nervosa, there have been no previous definitive placebo-controlled studies evaluating the effectiveness of oral contraceptive treatment on bone mineral density in pediatric females with anorexia nervosa. This is a randomized (patients are assigned different treatments based on chance), multicenter, double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), placebo-controlled study to evaluate the bone mineral density in pediatric patients with anorexia nervosa following treatment with norgestimate/ethinyl estradiol or placebo for 13 consecutive 28-day cycles. Norgestimate/Ethinyl Estradiol is packaged in a 28-day blistercard. Each tablet contains the following:

a) Days 1-7 0.180 mg norgestimate/0.035 mg ethinyl estradiol b) Days 8-14 0.215 mg norgestimate/0.035 mg ethinyl estradiol c) Days 15-21 0.250 mg norgestimate/0.035 mg ethinyl estradiol d) Days 22-28 inactive tablets;One tablet is to be taken once daily by mouth. After 28 days, the next cycle is started the following day without interruption. Color-matched placebo tablets are identically pack

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a monthly period
* health status consistent with anorexia nervosa
* meet the modified DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) guideline for anorexia nervosa
* must discontinue the following prior to Baseline visit: hormonal contraceptives for 3 months
* hormonal intrauterine devices (IUDs) for 1 month
* NORPLANT for 3 months
* DepoProvera and other depot hormone injections, for 6 months
* Lupron, Lupron Depot 3.75 mg and 7.5 mg, Synarel, Zoladex, Cetrotide for 3 months
* Lupron Depot 11.25 mg, 15 mg, 22.5 mg, 30 mg for 6 months
* non-smoker or smoking <= 15 cigarettes per day
* must agree to use reliable non-hormonal alternate method of birth control during the study

Exclusion Criteria:

* History or presence of disorders commonly accepted as contraindications to steroid hormonal therapy including but not limited to the following - active or history of deep vein thrombophlebitis or thromboembolytic disorders or hypercoagulation disorders, cerebral vascular or coronary artery disease, uncontrolled hypertension, or migraines with focal aura, benign or malignant liver tumor which developed during the use of oral contraceptives or estrogen-containing products, known or suspected carcinoma of any body system, diabetes mellitus with vascular involvement
* recent history of alcohol or substance abuse
* patients with primary amenorrhea (abnormal suppression or absence of menstruation) who in the opinion of the physician, are not appropriate candidates for hormonal therapy (eg, have not grown to an acceptable adult height)
* subjects who are suicidal
* patients who have received any experimental drug and/or used any experimental device within 30 days before the start of the study.

Max Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
The change in total lumbar spine (L1-L4) bone mineral density from baseline to Cycle 6 (Visit 6).

SECONDARY OUTCOMES:
The percent change in total lumbar spine BMD from baseline to Cycle 6. The change and percent change in total lumbar spine BMD from baseline to Cycle 13. The change and percent change in total hip BMD from baseline to Cycle 6 and Cycle 13.

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Result] Strokosch GR, Friedman AJ, Wu SC, Kamin M. Effects of an oral contraceptive (norgestimate/ethinyl estradiol) on bone mineral density in adolescent females with anorexia nervosa: a double-blind, placebo-controlled study. J Adolesc Health. 2006 Dec;39(6):819-27. doi: 10.1016/j.jadohealth.2006.09.010. PMID 17116511